CLINICAL TRIAL: NCT02866513
Title: Incidence of High Levels of Transpulmonary Pressure During the Use of Airway Pressure Release Ventilation.
Brief Title: Transpulmonary Pressure and Airway Pressure Release Ventilation (APRV).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-19
Record Dates: First submitted 2016-08-02; First posted 2016-08-15 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2016-08

CONDITIONS: Patient Mechanically Ventilated With APRV Mode

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient mechanically ventilated with APRV mode (Other)
  Interventions: Other: evaluate the variations of transpulmonary pressure during the use of APRV by clinicians.

INTERVENTIONS:
Other: evaluate the variations of transpulmonary pressure during the use of APRV by clinicians.

SUMMARY:
Mechanical ventilation can induce pulmonary lesions called ventilator induced lung injury (VILI). High levels of Transpulmonary pressure is one of the most important mechanism of VILI during the use of mechanical ventilation. The use of bilevel pressure ventilator modes like APRV could generate high levels of transpulmonary pressure.

The aim of this study is to evaluate the variations of transpulmonary pressure during the use of APRV by clinicians

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patient mechanically ventilated for more than 48 H for acute respiratory failure
* Decision to use of the APRV mode by clinicians in charge of the patient

Exclusion Criteria:

- Contraindication for the use of a nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Transpulmonary pressure | 24 hours
  Measurement of transpulmonary pressure needs the measurement of oesophageal pressure with a specific nasogastric tube. This measurement is now available in routine in few mechanical ventilators in intensive care units (eg: AVEA Ventilator. Vyasys HealthCare). Transpulmonary pressure is the difference between airway pressure and oesophageal pressure and it is now easy to obtain and monitor at the bedside with these ventilators. It is also possible to record the value furthermore than 24 hours.

SECONDARY OUTCOMES:
Maximal value of transpulmonary pressure | 24 hours
  Value of tidal volume > 8 ml/kg

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille hôpital de la Timone, Marseille, France